CLINICAL TRIAL: NCT06940544
Title: Uppsala Self-SCREENing of Heart Failure Study
Acronym: U-SCREEN-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2022-06248-01
Record Dates: First submitted 2025-03-17; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; Home-based screening; Point-of-care testing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCREENING Arm (Experimental): Home-Based HF Screening with NTproBNP and AI-Assisted Echocardiography
  Interventions: Diagnostic Test: Stepwise Multimodal Home-Based HF Screening
- CONTROL Arm (No Intervention): Usual Care Without Systematic HF Screening

INTERVENTIONS:
Diagnostic Test: Stepwise Multimodal Home-Based HF Screening — The Stepwise Multimodal Home-Based HF Screening intervention involves a targeted community outreach program to identify undiagnosed heart failure (HF) in high-risk individuals. Participants randomized to the intervention arm (ACTIVE) are asked to self-collect dried blood spots for NTproBNP analysis. Those with elevated NTproBNP (≥125 pg/ml) in the dried blood spots are summoned to the study clinic and undergo confirmatory point-of-care NTproBNP testing and an AI-enabled echocardiogram, with the aim to confirm or rule out heart failure.
  Arms: SCREENING Arm

SUMMARY:
The goal of this clinical trial is to investigate whether a stepwise multimodal home-based screening strategy with rapid point-of-care testing can detect undiagnosed heart failure (HF) in high-risk patients compared to usual care. The study also aims to understand the impact of earlier HF diagnosis on treatment initiation, clinical outcomes, symptoms, functional capacity, health-related quality of life, healthcare utilization, and costs.

The main questions it aims to answer are:

Does a home-based screening strategy increase the diagnosis of HF within 6 months compared to usual care?

Does earlier diagnosis lead to more patients receiving guideline-directed medical therapy (GDMT) for HF with reduced ejection fraction (HFrEF) within 6 months?

What is the impact of this screening strategy on HF hospitalizations, mortality, functional capacity, health-related quality of life, and healthcare costs over 1, 2, and 5 years?

Researchers will compare a stepwise multimodal home-based screening strategy to usual care to determine if the screening strategy leads to earlier HF diagnosis and improved patient outcomes.

Participants will:

Provide dried blood spot samples for NTproBNP analysis by mail.

If NTproBNP is elevated (≥125 pg/ml), undergo point-of-care NTproBNP testing and an AI-enabled echocardiogram.

Be followed for up to 5 years through healthcare databases and self-reported symptom monitoring to track HF diagnosis, treatment initiation, clinical outcomes, and healthcare utilization.

The study will randomize 500 high-risk participants in a 1:1 ratio to either the ACTIVE arm (home-based screening) or the CONTROL arm (usual care). Participants with known HF are excluded.

The primary outcome is the diagnosis of HF within 6 months. Secondary outcomes include the diagnosis of HFrEF and initiation of GDMT within 6 months. Exploratory outcomes will assess long-term clinical outcomes (HF hospitalizations and death), functional capacity, quality of life, and cost-effectiveness at 1, 2, and 5 years.

This investigator-initiated trial is part of the international SYMPHONY study and is coordinated from Uppsala University and Uppsala University Hospital, Sweden. The study will use healthcare databases, registries, and digital resources for comprehensive outcome capture. The first patient visit is scheduled for February 1, 2023, with follow-up extending to August 2026 for the primary outcome and up to 5 years for exploratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

Age ≥40 years, and at least one of the following symptoms of HF, and at least two risk factors for HF:

Symptoms

* Dyspnoea on exertion
* Dyspnoea at rest
* Orthopnoea
* Paroxysmal nocturnal dyspnoea
* Reduced exercise tolerance, increased time to recover after exercise
* Fatigue, tiredness
* Ankle swelling

Risk factors

* Diabetes (type 1 or type 2)
* Coronary artery disease (myocardial infarction or coronary artery bypass grafting or percutaneous coronary intervention)
* Persistent or permanent atrial fibrillation (not paroxysmal atrial fibrillation)
* Previous ischemic or embolic stroke
* Peripheral arterial disease (previous surgical or percutaneous revascularisation)
* Chronic kidney disease
* Regular loop diuretic use (any dose at any dosing interval) for >30 days
* COPD (diagnosis by respiratory physician, radiological emphysema or treatment with advocated COPD therapy)

Exclusion Criteria:

* Previous diagnosis of HF
* Previous renal replacement therapy
* Inability to comply with study procedures or provide informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Detection of undiagnosed heart failure (HF) in high-risk patients. | Within 6 months.
  Diagnosis of HF; HF is defined as either:
  1. an outpatient diagnosis of heart failure according to the ESC 2021 Heart Failure Guidelines,
  2. outpatient heart failure visit,
  3. an urgent heart failure visit, or
  4. a heart failure hospitalisation.

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala Akademiska Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of certain IPD may be prohibited for ethical reasons.

REFERENCES:
- [Background] McGrady M, Krum H, Carrington MJ, Stewart S, Zeitz C, Lee GA, Marwick TH, Haluska BA, Brown A. Heart failure, ventricular dysfunction and risk factor prevalence in Australian Aboriginal peoples: the Heart of the Heart Study. Heart. 2012 Nov;98(21):1562-7. doi: 10.1136/heartjnl-2012-302229. Epub 2012 Aug 11. PMID 22888160
- [Background] Packer M. Do most patients with obesity or type 2 diabetes, and atrial fibrillation, also have undiagnosed heart failure? A critical conceptual framework for understanding mechanisms and improving diagnosis and treatment. Eur J Heart Fail. 2020 Feb;22(2):214-227. doi: 10.1002/ejhf.1646. Epub 2019 Dec 17. PMID 31849132
- [Background] Tromp J, Seekings PJ, Hung CL, Iversen MB, Frost MJ, Ouwerkerk W, Jiang Z, Eisenhaber F, Goh RSM, Zhao H, Huang W, Ling LH, Sim D, Cozzone P, Richards AM, Lee HK, Solomon SD, Lam CSP, Ezekowitz JA. Automated interpretation of systolic and diastolic function on the echocardiogram: a multicohort study. Lancet Digit Health. 2022 Jan;4(1):e46-e54. doi: 10.1016/S2589-7500(21)00235-1. Epub 2021 Dec 1. PMID 34863649
- [Background] Jorgensen B, Bertsch T, Broker HJ, Schafer M, Chapelle JP, Gadisseur R, Cowie MR, Dikkeschei B, Gurr E, Hayen W, Hafner G, Stiegler Y, Schonherr HR, Strasser RH, Weidtmann B, Folkerts H, Zugck C, Hofmann K, Zerback R. Multicentre evaluation of a second generation point-of-care assay with an extended range for the determination of N-terminal pro-brain natriuretic peptide. Clin Lab. 2012;58(5-6):515-25. PMID 22783583
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Sundstrom J, Lind L, Nowrouzi S, Lytsy P, Marttala K, Ekman I, Ohagen P, Ostlund O. The Precision HYpertenSIon Care (PHYSIC) study: a double-blind, randomized, repeated cross-over study. Ups J Med Sci. 2019 Jan;124(1):51-58. doi: 10.1080/03009734.2018.1498958. Epub 2018 Sep 28. PMID 30265168
- [Background] Goldman L, Hashimoto B, Cook EF, Loscalzo A. Comparative reproducibility and validity of systems for assessing cardiovascular functional class: advantages of a new specific activity scale. Circulation. 1981 Dec;64(6):1227-34. doi: 10.1161/01.cir.64.6.1227. PMID 7296795
- [Background] Homar V, Mirosevic S, Svab I, Lainscak M. Natriuretic peptides for heart failure screening in nursing homes: a systematic review. Heart Fail Rev. 2021 Sep;26(5):1131-1140. doi: 10.1007/s10741-020-09944-w. PMID 32200491
- [Background] Ontario Health (Quality). Use of B-Type Natriuretic Peptide (BNP) and N-Terminal proBNP (NT-proBNP) as Diagnostic Tests in Adults With Suspected Heart Failure: A Health Technology Assessment. Ont Health Technol Assess Ser. 2021 May 6;21(2):1-125. eCollection 2021. PMID 34055110
- [Background] Mant J, Doust J, Roalfe A, Barton P, Cowie MR, Glasziou P, Mant D, McManus RJ, Holder R, Deeks J, Fletcher K, Qume M, Sohanpal S, Sanders S, Hobbs FD. Systematic review and individual patient data meta-analysis of diagnosis of heart failure, with modelling of implications of different diagnostic strategies in primary care. Health Technol Assess. 2009 Jul;13(32):1-207, iii. doi: 10.3310/hta13320. PMID 19586584
- [Background] Thorstensen A, Dalen H, Amundsen BH, Aase SA, Stoylen A. Reproducibility in echocardiographic assessment of the left ventricular global and regional function, the HUNT study. Eur J Echocardiogr. 2010 Mar;11(2):149-56. doi: 10.1093/ejechocard/jep188. Epub 2009 Dec 3. PMID 19959533
- [Background] Nagueh SF, Abraham TP, Aurigemma GP, Bax JJ, Beladan C, Browning A, Chamsi-Pasha MA, Delgado V, Derumeaux G, Dolci G, Donal E, Edvardsen T, El Tallawi KC, Ernande L, Esposito R, Flachskampf FA, Galderisi M, Gentry J, Goldstein SA, Harb SC, Hubert A, Hung J, Klein AL, Lancellotti P, Mahmood RZ, Marino P, Popescu BA, Previato M, Sanghai SR, Smiseth OA, Xu J; for Diastolic Function Assessment Collaborators. Interobserver Variability in Applying American Society of Echocardiography/European Association of Cardiovascular Imaging 2016 Guidelines for Estimation of Left Ventricular Filling Pressure. Circ Cardiovasc Imaging. 2019 Dec;12(1):e008122. doi: 10.1161/CIRCIMAGING.118.008122. PMID 30632389
- [Background] Ezekowitz JA, Kaul P, Bakal JA, Quan H, McAlister FA. Trends in heart failure care: has the incident diagnosis of heart failure shifted from the hospital to the emergency department and outpatient clinics? Eur J Heart Fail. 2011 Feb;13(2):142-7. doi: 10.1093/eurjhf/hfq185. Epub 2010 Oct 19. PMID 20959343
- [Background] Conrad N, Judge A, Canoy D, Tran J, O'Donnell J, Nazarzadeh M, Salimi-Khorshidi G, Hobbs FDR, Cleland JG, McMurray JJV, Rahimi K. Diagnostic tests, drug prescriptions, and follow-up patterns after incident heart failure: A cohort study of 93,000 UK patients. PLoS Med. 2019 May 21;16(5):e1002805. doi: 10.1371/journal.pmed.1002805. eCollection 2019 May. PMID 31112552
- [Background] Koudstaal S, Pujades-Rodriguez M, Denaxas S, Gho JMIH, Shah AD, Yu N, Patel RS, Gale CP, Hoes AW, Cleland JG, Asselbergs FW, Hemingway H. Prognostic burden of heart failure recorded in primary care, acute hospital admissions, or both: a population-based linked electronic health record cohort study in 2.1 million people. Eur J Heart Fail. 2017 Sep;19(9):1119-1127. doi: 10.1002/ejhf.709. Epub 2016 Dec 23. PMID 28008698
- [Background] van Riet EE, Hoes AW, Limburg A, Landman MA, van der Hoeven H, Rutten FH. Prevalence of unrecognized heart failure in older persons with shortness of breath on exertion. Eur J Heart Fail. 2014 Jul;16(7):772-7. doi: 10.1002/ejhf.110. Epub 2014 May 26. PMID 24863953
- [Background] Bottle A, Kim D, Aylin P, Cowie MR, Majeed A, Hayhoe B. Routes to diagnosis of heart failure: observational study using linked data in England. Heart. 2018 Apr;104(7):600-605. doi: 10.1136/heartjnl-2017-312183. Epub 2017 Oct 5. PMID 28982720
- [Background] Braunwald E. The war against heart failure: the Lancet lecture. Lancet. 2015 Feb 28;385(9970):812-24. doi: 10.1016/S0140-6736(14)61889-4. Epub 2014 Nov 16. PMID 25467564
- [Background] Virani SS, Alonso A, Aparicio HJ, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Cheng S, Delling FN, Elkind MSV, Evenson KR, Ferguson JF, Gupta DK, Khan SS, Kissela BM, Knutson KL, Lee CD, Lewis TT, Liu J, Loop MS, Lutsey PL, Ma J, Mackey J, Martin SS, Matchar DB, Mussolino ME, Navaneethan SD, Perak AM, Roth GA, Samad Z, Satou GM, Schroeder EB, Shah SH, Shay CM, Stokes A, VanWagner LB, Wang NY, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2021 Update: A Report From the American Heart Association. Circulation. 2021 Feb 23;143(8):e254-e743. doi: 10.1161/CIR.0000000000000950. Epub 2021 Jan 27. PMID 33501848
- [Background] Cook C, Cole G, Asaria P, Jabbour R, Francis DP. The annual global economic burden of heart failure. Int J Cardiol. 2014 Feb 15;171(3):368-76. doi: 10.1016/j.ijcard.2013.12.028. Epub 2013 Dec 22. PMID 24398230
- [Background] Bragazzi NL, Zhong W, Shu J, Abu Much A, Lotan D, Grupper A, Younis A, Dai H. Burden of heart failure and underlying causes in 195 countries and territories from 1990 to 2017. Eur J Prev Cardiol. 2021 Dec 29;28(15):1682-1690. doi: 10.1093/eurjpc/zwaa147. PMID 33571994
- See also: Digital consent platform with current version of participant information, and possibility to consent to the study during the recruitment period — https://u-screen-hf.minforskning.se